CLINICAL TRIAL: NCT00318019
Title: The Effect of OPC Factor on Energy Levels in Healthy Individuals Aged 45-65: A Randomized Controlled Trial
Brief Title: Effect of OPC Factor on Energy Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 804315
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Energy; Energy Level

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- OPC Factor(TM) (Experimental)
  Interventions: Dietary Supplement: OPC Factor(TM)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: OPC Factor(TM) — Evervescent poweder containing oligomeric proanthocyanidins (OPCs)and other nutrients.
  Arms: OPC Factor(TM)
Other: Placebo — Effervescent powder similar in taste and appearance to the intervention but without the OPCs and nutrients.
  Arms: Placebo

SUMMARY:
In this study the food supplement OPC Factor will be tested to determine its effectiveness for increasing energy levels in healthy people aged 45-65 when compared to a placebo. All subjects will receive both active product and placebo at some time during the study. The study is nine weeks in duration. It involves three visits, taking an effervescent powder in water twice a day, and answering 24 multiple choice questions once a week. Subjects who complete the study can elect to receive a two month supply of the study product free of charge.

DETAILED DESCRIPTION:
OPC Factor, a food supplement which contains grape seed extract, pine bark extract,vitamins and minerals, has shown during clinical observation the effect of raising energy levels in people aged 45-65. It is believed that the mechanism of action is based on enhanced production of ATP by mitochondria.

In this study subjects will be assigned by chance to either the active product group or the placebo group. Subjects will take the product for three weeks. Then there will be a two week wash out period followed by subjects being crossed over to the other group for a three week period. Subjects, assessors, and health providers will be masked as to who is in the active product group and who is in the placebo group. Subjects will meet with the primary investigator three times during the study, will fill out very short questions once a week, and receive phone calls once a week from study personnel.

This study is a randomized, placebo controlled, triple-blinded, cross-over study that tests the hypothesis that OPC Factor produces a response rate of 70% in the active product phase versus a 30% response rate during the placebo phase. A response is defined as at least a 20% absolute increase on the Energy subscale of the Activation-Deactivation Adjective Check List.

ELIGIBILITY:
Inclusion Criteria:

1. 45 to 65 years of age at the time of recruitment
2. Healthy -- see exclusion criteria
3. There is the possibility of at least a 20% absolute increase in the subject's energy subscale score of the Activation-Deactivation Adjective Checklist (AD ACL). For the purpose of meeting the inclusion criteria, the subject fills out the AD ACL with the following instructions: "Each of the words below describes feelings or moods. Please circle the rating next to each word that best describes your feelings during the past month. These instructions are different from the instructions used when the study endpoints are being measured so as to be consistent with the way the questionnaire was validated."

Exclusion Criteria:

1. Any major medical or mental illness (including a history of bipolar disorder, borderline personality disorder, and schizophrenia)
2. Medical diseases known to be associated with fatigue but not limited to:

   * AIDS
   * Anemia
   * Cancer or history of cancer (excluding basal cell carcinoma of the skin)
   * Chronic fatigue syndrome
   * Congestive heart failure
   * Chronic obstructive pulmonary disease (COPD)
   * Depression
   * Diabetes
   * Drug/alcohol dependence
   * Fibromyalgia
   * Hypertension that is uncontrolled or difficult to control
   * Hypothyroidism
3. Subjects taking the following medical therapies:

   * Beta-blocking medications
   * Human growth hormone
   * Testosterone
   * Warfarin
4. Subjects taking the following complementary and alternative medicine (CAM) products:

   * Feverfew
   * Garlic supplements
   * Ginseng
   * Red clover
5. Women who have not gone through menopause - those women who have had one or more menstrual periods in the 12 months prior to the enrollment in the study
6. The subject's score on the energy subscale of the AD ACL is at a level that precludes at least a 20% absolute increase of that score.
7. Subjects who are unable to make their own decisions regarding informed consent
8. Those subjects who have taken any of the medical therapies or CAM products listed but are no longer taking them are eligible to participate provided no other exclusion criteria are present and the subjects have not taken those therapies or products in the six months prior to enrollment.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Energy subscore on the Activation-Deactivation Adjective Check List | Nine weeks

SECONDARY OUTCOMES:
Four global change questions | Nine weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J LaRiccia, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States